CLINICAL TRIAL: NCT05449678
Title: The LATTITUDE Study - Low Carbohydrate Diet and Automated Insulin Delivery System for Type 1 Diabetes
Brief Title: Low cArbohydraTe dIeT and aUtomated Insulin Delivery System for Type 1 DiabetEs
Acronym: LATITUDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1182
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet (No Intervention): Usual diet (45% of daily energy intake from CHO)
- Low carb diet (Experimental): Low-carb diet (25% of daily energy intake from CHO)
  Interventions: Behavioral: Low-carb diet

INTERVENTIONS:
Behavioral: Low-carb diet — A close nutritional follow-up will take place with a qualified nutritionist to adapt the participants' usual diet to their assignment diet. This is not a strict diet to follow or a ketogenic diet. Nutritional modifications will be based on the participants' usual diet to improve adherence (personalized follow-up).
  Arms: Low carb diet

SUMMARY:
This is a randomized, controlled study in people living with type 1 diabetes using an automated insulin delivery (AID) system. Participants will be assigned to a control diet (45% carbohydrate) or a low carb diet (25% carbohydrate). The objective is to establish whether the low-carb diet improves time to glycemic targets at 3 months and whether the diet is realistically maintained at 1 year in patients using an AID-DIY system.

DETAILED DESCRIPTION:
Problems: Despite significant technological and treatment advances for people living with with type 1 diabetes (PWT1D), time in optimal glycemic targets remains difficult to achieve (between 4.0 and 10.0 mmol/L). On the other hand, there is increasing interest in low-carbohydrate diets in the general population (often for weight control), but also in people with diabetes, to help achieve glycemic control (associated with an increase in time in range (TIR).

Automated insulin delivery (AID) systems, including a continuous glucose monitor (CGM) coupled to an insulin pump with an integrated infusion algorithm, increase TIR by approximately 2 hours per day and reduce time in hypoglycemia by 30 minutes, compared to conventional treatments for type 1 diabetes. However, maintaining an optimal TIR remains a significant challenge for PWT1D, despite the increasing use of this technology.

AID systems in combination with a low-carbohydrate diet to optimize TIR have not been studied.

Objectives: To investigate whether low-carb diets improve glucose management and the feasibility of adopting low-carb diets among PWT1D using an AID.

Methods: This is a 12-month prospective, open-label, randomized, controlled study in adults living with type 1 diabetes, with the first 12 weeks as the main study phase and the rest as the extended study phase.

1. Admission period (2-4 weeks): Optimization of insulin doses, validation of carbohydrate calculations and maintenance of usual diet.
2. Main study period (3 months): Study assignment diet (low carbohydrate or usual).
3. Extensive study phase (9 months): Maintenance of assignment diet (if possible) with less frequent visits (observation period).

Hypothesis: The low-carb diet would increase the TIR% (primary outcome) by a mean of 8% (SD 8) compared with the usual diet. Power calculation: Using mean 8% (SD 8), that 38 adults (19 for each group) would provide 80% power at the 5% significance level to detect differences between the two interventions, after considering a 10% drop-out rate.

Full analysis set is defined as participants who have finished recruitment. Per-protocol set is defined as participants who have finished recruitment and have at least 70% of CGM data, at least 70% time in closed-loop mode and at least 4 full days of diet data during week 3-4. The efficiency analysis will be performed using the per-protocol set. The safety analysis will be performed using the full analysis set.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old
2. Duration of T1D or latent autoimmune diabetes in adults (LADA) ≥ 12 months
3. On automated insulin delivery system for ≥ 3 months
4. Own a smartphone or tablet to use the mobile application: Keenoa
5. Willing to share personal CGM data during the study period
6. Reporting daily food intake >3350 kJ (1200 kcal)
7. Time in closed-loop mode during run-in period > 70%

Exclusion Criteria:

1. Self-reported having a diet with < 35% energy from carb.
2. Seldom (<20% of scenario) or never count carbohydrate intake.
3. Self-reported clinically significant nephropathy (eGFR < 30 ml/min/1.73m2, planned or on dialysis or already followed by a nephrologist), or retinopathy (e.g., proliferative retinopathy with ongoing active treatment such as laser photocoagulation or planned surgery)
4. Recent (< 6 months) acute macrovascular event (e.g., acute coronary syndrome or cardiac surgery).
5. Self-reported significant liver disease (e.g. cirrhosis, active hepatitis, liver transplantation)
6. Self-reported uncontrolled thyroid disease (unless stable treatment for 8 weeks at inclusion with TSH within target range).
7. Self-reported one or more severe hypoglycemic episodes within two weeks of screening.
8. Self-reported one or more severe hyperglycemic episodes requiring hospitalization in the last 3 months.
9. Anticipated therapeutic change (including change of insulin type [switch to biosimilar is not considered as insulin change] and/or type of CGM sensor, insulin pump or AID between admission and end of the study.
10. To limit risk of interference for CGM accuracy: anticipated need to use acetaminophen during the study period at a dose above 1g every 6 hours and current or anticipated use of Hydroxyurea.
11. Plan to go abroad in a foreign country during the study period for a duration > 4 weeks.
12. Pregnancy (ongoing or current attempt to become pregnant).
13. Breastfeeding.
14. Using regular insulin (Entuzity U500, Novolin ge Toronto or Humulin R).
15. Current use of glucocorticoid medication (except low stable dose and inhaled steroids and stable adrenal insufficiency treatment e.g., Cortef®).
16. Current use of agents affecting gastric emptying (Motilium®, Victoza®, Ozempic®, Trulicity®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, Prandase®, DPP-4 inhibitors) unless at a stable dose for 3 months and without anticipated change during the study.
17. Current use of SGLT-2 inhibitors unless at a stable dose for at least 3 months, without anticipated change during the study and appropriate ketone testing is performed.
18. Other serious medical illnesses which likely interfere with study participation or with the ability to complete the study by the judgment of the investigator.
19. In the opinion of the investigator, a participant who is unable or unwilling to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) | 12 weeks
  The comparison between low-carb diet and usual diet regarding percentage of time of glucose levels spent between 3.9 and 10.0 mmol/L (TIR%) based on sensor glucose value during week 11 and 12 (24-hour).

SECONDARY OUTCOMES:
Adherence | 1 year
  Adherence to the prescribed diet (average % CHO intakes/day; number of days with +/- 5% CHO of prescribed diet; % meals following +/-5% targeted CHO)

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, MD, PhD, Study Director — IRCM

IPD SHARING:
Plan to Share IPD: No